CLINICAL TRIAL: NCT00207116
Title: An Exploratory Pharmacogenomic Study of Monotherapy Erbitux in Subjects With Metastatic Non Small Cell Lung Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-065; NCT00118118 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis
Keywords: Metastatic Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Cetuximab

ARMS (1):
- A (Experimental)
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — IV solution, IV, 400 mg/m2 initial dose followed by weekly doses of 250 mg/m2, Weekly, until disease progression.
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to predict responses to Erbitux as a single agent in patients with Non Small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease tumor available for biopsies
* Life expectancy of at least 3 months

Exclusion Criteria:

* Known or documented brain metastases prior to Cetuximab therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Prediction of response to Erbitux with non small cell lung cancer

SECONDARY OUTCOMES:
Radiographic Response

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Local Institution, Newark, Delaware, United States